CLINICAL TRIAL: NCT00216697
Title: An Extension or Re-Treatment Study of Bortezomib to Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: An Extension Study to Provide Bortezomib to Patients With Relapsed or Refractory Multiple Myeloma Who Previously Participated in a Bortezomib Phase I/II Study and Who May Benefit From Re-Treatment With or Continuation of Bortezomib Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004843
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Proteasome inhibitor; Ubiquitin; Boronic acids; Bortezomib
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
One purpose of this study is to evaluate the effectiveness and safety in long term treatment for patients who completed preceding phase I/II study. The other purpose is to evaluate the effectiveness and safety of patients who are re-treated with this drug in recommended dose.

DETAILED DESCRIPTION:
Multiple myeloma is a kind of malignant disease in the organ which produce blood cells such as bone marrow. It has poor prognosis, especially in patients who are relapsed repeatedly. Effective treatment is strongly expected in such relapsed patients in Japan. This is a open label multiple center study to evaluate the effectiveness and safety of bortezomib. This study is an extension or re-treatment study for patients who were administered with bortezomib in preceding Phase I/II study. For extension treatment, the same dose of the previous study will be administered into a vein as a bolus twice weekly followed by a 10-day rest (3-week cycle). For re-treatment, a recommended dose determined in Phase I/II study will be administered in 3-week cycle.

ELIGIBILITY:
Inclusion Criteria:

* Complete 6 cycles treatment in preceding phase I/II study
* response (CR, PR, MR or NC) was obtained in 6 cycles treatment during the preceding phase I/II study and investigator considers that the patient is expected to have benefit such as antitumor effect, pain relief or improvement of performance state
* Patients who did not have Grade >=3 non-hematologic toxicity or Grade 4 hematologic toxicity during the preceding phase I/II study or extension treatment of this study
* Investigator considers that the patient is expected to have benefit of this drug such as antitumor effect, pain relief or improvement of performance state.

Exclusion Criteria:

* Patient is known to be HBs antigen positive, HCV antibody positive or HIV antibody positive (check is required for patients who received blood product during phase I/II study)
* Patients who receive G-CSF product or blood transfusion within 7 days before the start of treatment
* Disease progress was observed during the phase I/II or this study when patients receive recommended dose
* Patients who suffer Grade >=2 peripheral neuropathy or Grade >=2 neuropathic pain
* Patient has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, acute ischemia or active conduction system abnormalities.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-03; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
No. of patients who had adverse events, incidence and severity of adverse events, and relationship to the study drug. Overall response rate (Complete Remission + Partial Remission). Response will be evaluated by independent review committee.

SECONDARY OUTCOMES:
TTP (Time To Progression), survival time, time to response and duration of response. For re-treatment patients, survival time from the previous study drug treatment and response rate from the start of re-treatment will be also evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.

REFERENCES:
- See also: A Continuous Administration or Readministration Study JNJ-26866138 (bortezomib) in Patients with Relapsed or Refractory Multiple Myeloma — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=404&filename=CR004843_CSR.pdf